CLINICAL TRIAL: NCT04309994
Title: Combined Use of a Novel Cardioplegic Formula With MPS® Versus Cardioplexol ® in Urgent Isolated CABG Using MiECC in Patients With Recent Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-02383; ch20Reuthebuch
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Heart Attack; Cardioplegia Solution Adverse Reaction; Coronary Artery Bypass Grafting (CABG)
Keywords: heart attack; cardioplegia solution; Minimal extracorporeal circulation system (MiECC); Myocardial protection system (MPS); Coronary artery bypass grafting (CABG)
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: bypass surgery with blood cardioplegia by means of MPS
  Interventions: Other: Myocardial protection system (MPS)
- Active Comparator: bypass surgery with blood cardioplegia by means of Cardioplexol ®
  Interventions: Other: Cardioplexol

INTERVENTIONS:
Other: Myocardial protection system (MPS) — cardioplegia solution, A separate pumpsystem by which Blood cardioplegia with individually composable additives as cardioplegia solution can be used
  Groups: Experimental
Other: Cardioplexol — cardioplegia solution
  Groups: Active Comparator

SUMMARY:
The goal of this study is to compare the two cardioplegia solutions (blood cardioplegia by means of MPS ® vs. Cardioplexol ®) regarding perioperative outcome and with special attention to cardiac markers in patients with a recent heart attack.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent a CABG using MPS® or Cardioplexol ®
* Heart attack less than 7 days before surgery

Exclusion Criteria:

* use of other cardioplegia solution than Cardioplexol ® or MPS®
* other inventions than CABG
* explicit will of the patient that his data may not be used
* denied general consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients which underwent isolated CABG (coronary artery bypass grafting) using MiECC (Minimal extracorporeal circulation system) at the department of cardial surgery University Hospital Basel Switzerland
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
myocardial damage | patients with that received a coronary artery bypass grafting and that were treated (for approximately 15 days) at the University Hospital between February 2010 and January 2020 (data taken perioperative during hospital stay for CABG)
  Analyse cardiac biomarkers as indicators for myocardial damage: high sensitive troponin (Ths-TrT, ng/mL), creatine kinase (CK, in ng/mL) and creatine kinase-MB isoenzyme (CK-MB, in ng/mL)

SECONDARY OUTCOMES:
30 days Mortality | 30 days after CABG
  death after coronary artery bypass grafting
length of stay in the intensive care unit | perioperative during hospital stay for CABG (for approximately 15 days)
  duration of stay at intensive care unit
Number of participants with bleedings | perioperative during hospital stay for CABG (for approximately 15 days)
  bleeding complication after coronary artery bypass grafting
Number of participants with postoperative arrhythmia | perioperative during hospital stay for CABG (for approximately 15 days)
  rhythm disturbance after coronary artery bypass grafting

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Reuthebuch, Prof. Dr. med., Principal Investigator — Cardiac Surgery Clinic, University Hospital Basel
Locations (1):
- Cardiac Surgery Clinic University Hospital Basel, Basel, Switzerland